CLINICAL TRIAL: NCT01208558
Title: Whole Grain Versus no Grain With or Without Physiotherapy-promoted Exercise for Waist Loss
Brief Title: Grain Exercise Trial - Whole Grain Versus no Grain With or Without Physiotherapy-promoted Exercise for Waist Loss
Acronym: GET
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Principal Investigator, TJonsson, MD, PhD, Lund University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: LU2010/332
Record Dates: First submitted 2010-09-23; First posted 2010-09-24 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Abdominal Obesity; Cardiovascular Diseases; Diabetes Type 2; Hypertension; Overweight
Keywords: Blood pressure; Cereals; Diet Therapy; Dietary carbohydrates; Dietary fiber; Exercise Therapy; Food; Glucose intolerance; Lifestyle; Physiotherapy; Stroke; TIA; Waist circumference; Weight loss
MeSH Terms: conditions — Obesity, Abdominal; Cardiovascular Diseases; Diabetes Mellitus, Type 2; Hypertension; Overweight; Glucose Intolerance; Stroke; Weight Loss | interventions — Whole Grains; Physical Therapy Modalities; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Diet A and physiotherapy (Active Comparator): Behavioral: Diet A Prudent diet without grains. Written advice and 17-20 group sessions. Subjects are advised to avoid cereal grains. Apart from that, the recommendation is to follow Nordic Nutrition Recommendations (NNR) for overweight people, i.e. to eat much fruit, vegetables, fish, and to choose low-fat meat, and low-fat dairy products, and to avoid junk food and juice. In order to match carbohydrate intake between the arms, a high intake of potatoes, root vegetables, fruit and other carbohydrate-rich foods is recommended.
  Behavioral: Physiotherapy Twelve physiotherapy-led, charged, 2-hour sessions of structured group training for increased cardiorespiratory fitness. A pedometer sold at the start. Physical activity on prescription (FaR) at the end.
  Interventions: Behavioral: Diet A; Behavioral: Physiotherapy
- Diet B and physiotherapy (Active Comparator): Behavioral: Diet B Prudent diet with whole grains. Written advice and 17-20 group sessions. An exchange of regular cereal grains for whole grains is recommended. A daily intake of 7-8 portions of whole grain products is recommended, and a list of recommended cereal products (brands, names) is provided. Apart from that, the recommendation is identical to Diet A.
  Other Name: Whole grains Behavioral: Physiotherapy Twelve physiotherapy-led, charged, 2-hour sessions of structured group training for increased cardiorespiratory fitness. A pedometer sold at the start. Physical activity on prescription (FaR) at the end.
  Other Name: Exercise
  Interventions: Behavioral: Diet B; Behavioral: Physiotherapy
- Diet A only (Active Comparator): Behavioral: Diet A Prudent diet without grains. Written advice and 17-20 group sessions. Subjects are advised to avoid cereal grains as much as possible. Apart from that, the recommendation is to follow Nordic Nutrition Recommendations (NNR) for overweight people (www.slv.se; in Swedish), i.e. to eat much fruit, vegetables, fish, and to choose low-fat meat, and low-fat dairy products, and to avoid candy, ice cream, snacks, cakes, pastries, chocolate, potato chips, beer, soft drinks and juice. In order to match carbohydrate intake between the intervention arms, a high intake of potatoes, root vegetables, fruit and other carbohydrate-rich foods is recommended.
  Other Name: No grains
  Interventions: Behavioral: Diet A
- Diet B only (Active Comparator): Behavioral: Diet B Prudent diet with whole grains. Written advice and 17-20 group sessions. An exchange of regular cereal grains for whole grains is recommended. A daily intake of 7-8 portions of whole grain products is recommended, and a list of recommended cereal products (brands, names) is provided. Apart from that, the recommendation is identical to Diet A. The goal is that carbohydrate intake, as a proportion of total energy intake, should not differ between the groups.
  Other Name: Whole grains
  Interventions: Behavioral: Diet B
- Control (No Intervention): Only follow-up. No intervention.

INTERVENTIONS:
Behavioral: Diet A — Prudent diet without grains. Written advice and 17-20 group sessions. Subjects are advised to avoid cereal grains as much as possible. Apart from that, the recommendation is to follow Nordic Nutrition Recommendations (NNR) for overweight people (www.slv.se), i.e. to eat much fruit, vegetables, fish, and to choose low-fat meat, and low-fat dairy products, and to avoid candy, ice cream, snacks, cakes, pastries, chocolate, potato chips, beer, soft drinks and juice. In order to match carbohydrate intake between the intervention arms, a high intake of potatoes, root vegetables, fruit and other carbohydrate-rich foods is recommended.
  Guideline: 200-400 g of potatoes, 300-500 g of root crops, 400-600 g of vegetables, 200-300 g of beans, peas and corn, and 600 g of fruit and berries per day.
  Other Names: No grains
  Arms: Diet A and physiotherapy; Diet A only
Behavioral: Diet B — Prudent diet with whole grains. Written advice and 17-20 group sessions. An exchange of regular cereal grains for whole grains is recommended. A daily intake of 7-8 portions of whole grain products is recommended, and a list of recommended cereal products (brands, names) is provided. Apart from that, the recommendation is identical to Diet A: to follow Nordic Nutrition Recommendations (NNR) for overweight people (www.slv.se; in Swedish), i.e. to eat much fruit, vegetables, fish, and to choose low-fat meat, and low-fat dairy products, and to avoid candy, ice cream, snacks, cakes, pastries, chocolate, potato chips, beer, soft drinks and juice. The goal is that carbohydrate intake, as a proportion of total energy intake, should not differ between the groups.
  Other Names: Whole grains
  Arms: Diet B and physiotherapy; Diet B only
Behavioral: Physiotherapy — Twelve physiotherapy-led, charged, 2-hour sessions of structured group training for increased cardiorespiratory fitness. A pedometer sold at the start. Physical activity on prescription (FaR) at the end.
  Other Names: Exercise
  Arms: Diet A and physiotherapy; Diet B and physiotherapy

SUMMARY:
The main purpose of this 2-year lifestyle experiment for waist loss is twofold:

1. to compare whole grains and no grains as part of a healthy diet,
2. to determine if an 8-week exercise program, led by physiotherapists, is more efficient than brief counseling and follow-up.

People with abdominal overweight (≥84 cm in women and ≥98 cm in men) and at least one additional cardiovascular risk factor, (typically hypertension, diabetes type 2 or prior cardiovascular disease) are randomly assigned to receive Diet A or Diet B, with or without a structured exercise program at the department of physiotherapy, or to a control group receiving usual care. Diet A and B both include fruit, vegetables, fish, meat, and low-fat dairy products, and differ only in that Diet A recommends exchange of cereal grains for more potatoes, root vegetables, fruit and other carbohydrate-rich foods, while Diet B recommends exchange of regular cereal grains for whole grains. The primary outcome (most important follow-up variable) is change in waist circumference during 2 years. Secondary outcome measures include blood pressure, blood lipids, level of physical activity and, in subjects with diabetes, glycated hemoglobin and fasting blood sugar.

DETAILED DESCRIPTION:
This is a randomized controlled trial with 5 parallel groups of approximately equal size. Two hundred subjects with increased waist circumference (≥84 cm in women and ≥98 cm in men) and at least one additional cardiovascular risk factor will be included.

Four of the 5 groups will receive dietary advice (A or B) and 2 of them will be allocated to physiotherapy. A fifth control group will only receive usual care in addition to follow-up. Randomization will be performed by use of an internet-based random number generator from the School of Computer Science and Statistics, Trinity College, Dublin (www.random.org). randomly assigned to receive Diet A or Diet B, with or without a structured exercise program at the department of physiotherapy, or to a control group receiving usual care.

In addition to primary (waist loss) and secondary outcome measures as given below, a health questionnaire will be performed at baseline and after 12 and 24 months with questions about general health, self-reported quality of life, medication use, living habits, physical activity, nutrition, tobacco, alcohol, personal motivation and perceived ability to change lifestyle. Furthermore, serum creatinine will be measured at baseline, and after 3, 6, 12 and 24 months.

There are few randomized controlled trials comparing the effect of different lifestyle interventions on physical activity level or weight loss in overweight people at high risk of cardiovascular disease. There is no such study of the possible effect of a structured exercise program with group training led by physiotherapists, with the exception of rehabilitation programs after myocardial infarction. In addition, the possible unique effect of cereal grains on satiety and energy intake has not been addressed in randomized controlled trials. In two earlier studies in glucose intolerance and diabetes type 2, we have applied a dietary model (Paleolithic diet) based on root vegetables, fruit, vegetables, meat and fish, partly at the expense of cereal grains (Lindeberg et al., 2007; Jönsson et al., 2009). The results showed a more beneficial effect on waist circumference than from traditional dietary advice. In one of the studies in 29 overweight men with coronary heart disease and impaired glucose tolerance, the decrease of waist circumference was 2.7 cm greater (p=0,03) in the intervention group (-5.6 cm; 95% confidence interval [CI] -7.2;-3.9) than in the control group (-2.9, CI -4.8;-1.1) during 3 months of follow-up (Lindeberg et al., 2007). In the second study, where the same dietary model was applied in cross-over design among 13 subjects with diabetes type 2, waist circumference decreased 4 cm more (p=0,02) during the intervention diet than during the control diet (Jönsson et al., 2009). There is some evidence to suggest that cereal grains may interfere with leptin receptor activity in a way that could hypothetically suppress satiety (Jönsson et al., 2005; Kamikubo et al., 2008).

ELIGIBILITY:
Inclusion Criteria:

* increased waist circumference (≥84 cm in women and ≥98 cm in men)
* AND at least one additional cardiovascular risk factor: hypertension, diabetes type 2, prior coronary heart disease, prior stroke/TIA, peripheral arterial disease, impaired glucose tolerance, prior gestational diabetes, heredity or smoking

Exclusion Criteria:

* dependence on walking aids
* difficulty to understand Swedish (written or spoken)
* BMI >40 kg/m2
* cognitive impairment
* pronounced hearing loss
* aphasia
* continuous treatment with warfarin or prednisolone

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2010-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Change of waist circumference | 2 years
  Waist circumference (at elbow level) will be measured at baseline and after 3, 6, 12 and 24 months.

SECONDARY OUTCOMES:
Change of systolic and diastolic blood pressure | 2 years
  At baseline and after 3, 6, 12 and 24 months, sitting blood pressure will be measured twice at heart level with an automated device.
Change of body fat percentage | 2 years
  At baseline and after 12 and 24 months, total body fat percentage will be assessed by use of a Tanita hand-foot-BIA. Thickness of subcutaneous fat will be assessed by use of a Harpenden skinfold caliper at four sites (biceps, triceps, suprailiac and subscapular).
Change of plasma non-HDL cholesterol | 2 years
  Non-fasting plasma total and HDL cholesterol will be measured at baseline and after 3, 6, 12 and 24 months. HDL cholesterol will be subtracted from total cholesterol.
Change of physical activity level | 2 years
  A hip-mounted ActiGraph accelerometer will be worn daytime for six days at baseline and after 12 and 24 months for continuous monitoring of physical activity.
Change of glycated hemoglobin | 2 years
  Only in subjects with diabetes
Change of fasting blood sugar | 2 years
  Only in subjects with diabetes
Change of quantity and dosage of blood sugar-lowering drugs | 2 years
  All subjects will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Staffan Lindeberg, MD PhD, Study Chair — Center for Primary Health Care research, CRC, Lund University
Locations (1):
- Center for Primary Health Care Research, CRC, Lund University, Sweden, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lindeberg S, Jonsson T, Granfeldt Y, Borgstrand E, Soffman J, Sjostrom K, Ahren B. A Palaeolithic diet improves glucose tolerance more than a Mediterranean-like diet in individuals with ischaemic heart disease. Diabetologia. 2007 Sep;50(9):1795-1807. doi: 10.1007/s00125-007-0716-y. Epub 2007 Jun 22. PMID 17583796
- [Background] Jonsson T, Granfeldt Y, Ahren B, Branell UC, Palsson G, Hansson A, Soderstrom M, Lindeberg S. Beneficial effects of a Paleolithic diet on cardiovascular risk factors in type 2 diabetes: a randomized cross-over pilot study. Cardiovasc Diabetol. 2009 Jul 16;8:35. doi: 10.1186/1475-2840-8-35. PMID 19604407
- [Background] Kamikubo Y, Dellas C, Loskutoff DJ, Quigley JP, Ruggeri ZM. Contribution of leptin receptor N-linked glycans to leptin binding. Biochem J. 2008 Mar 15;410(3):595-604. doi: 10.1042/BJ20071137. PMID 17983356
- [Background] Jonsson T, Olsson S, Ahren B, Bog-Hansen TC, Dole A, Lindeberg S. Agrarian diet and diseases of affluence--do evolutionary novel dietary lectins cause leptin resistance? BMC Endocr Disord. 2005 Dec 10;5:10. doi: 10.1186/1472-6823-5-10. PMID 16336696
- [Derived] Rydhog B, Carrera-Bastos P, Granfeldt Y, Sundquist K, Jonsson T. Paleolithic diet fraction and score in post hoc data analysis of a randomized controlled trial with lifestyle interventions for abdominal obesity. BMC Nutr. 2025 Oct 2;11(1):180. doi: 10.1186/s40795-025-01165-4. PMID 41039470